CLINICAL TRIAL: NCT00040807
Title: Phase II Trial Of Weekly Irinotecan And Docetaxel In Recurrent Or Metastatic Head And Neck Carcinoma
Brief Title: Irinotecan and Docetaxel in Treating Patients With Metastatic or Locally Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069408; ECOG-E3301
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of irinotecan and docetaxel in treating patients who have metastatic or locally recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with metastatic or locally recurrent head and neck cancer treated with irinotecan and docetaxel.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Correlate angiogenesis markers and cyclooxygenase-2 expression with response and survival in patients treated with this regimen.
* Correlate UGT1A1 genotype with the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (no prior chemotherapy for locally recurrent or metastatic disease or more than 6 months since prior chemotherapy as primary therapy vs 1 prior chemotherapy regimen for locally recurrent or metastatic disease or less than 6 months since prior chemotherapy as primary therapy).

Patients receive docetaxel IV over 60 minutes followed by irinotecan IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 32-72 patients (16-36 per stratum) will be accrued for this study within 6-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma of the head and neck

  * Squamous cell carcinoma
  * No WHO grade II or III nasopharyngeal carcinoma (well-differentiated nasopharyngeal carcinoma allowed)
* Metastatic or locally recurrent disease considered to be incurable by locoregional therapy
* Unidimensionally measurable disease outside previously irradiated field unless documented progressive disease or histologically confirmed residual carcinoma at least 8 weeks after completion of radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST and ALT less than 2.5 times upper limit of normal (ULN) and alkaline phosphatase normal OR
* Alkaline phosphatase less than 4 times ULN and AST and ALT normal

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* No pre-existing grade 2 or greater peripheral neuropathy
* No other concurrent medical condition that would preclude study participation
* No hypersensitivity to drugs formulated with Polysorbate 80
* No other malignancy within the past 3 years except curatively treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior biologic therapy
* Any number of prior biologic therapies (e.g., chimeric antibodies or kinase inhibitors) allowed
* No concurrent filgrastim (G-CSF)

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No prior docetaxel or irinotecan
* No more than 1 prior chemotherapy regimen for recurrent or metastatic disease

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for recurrent or metastatic disease and recovered

Surgery:

* Recovered from prior surgery

Other:

* No concurrent antiepileptics
* No concurrent cyclosporine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11-19 (Actual); Primary Completion 2005-04 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (43):
- United States (43):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Denver Rose, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Argiris A, Buchanan A, Brockstein B, Kolesar J, Ghebremichael M, Pins M, Hahn K, Axelrod R, Forastiere A. Docetaxel and irinotecan in recurrent or metastatic head and neck cancer: a phase 2 trial of the Eastern Cooperative Oncology Group. Cancer. 2009 Oct 1;115(19):4504-13. doi: 10.1002/cncr.24528. PMID 19634157